CLINICAL TRIAL: NCT03532789
Title: Clinical Evaluation of Herbal Patch for Overactive Bladder Patients
Brief Title: Herbal Patch for Overactive Bladder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: En Chu Kong Hospital (Other)
Responsible Party: Principal Investigator, LIH-LIAN Chen, Attending physician of department of Traditional Chinese medicine, En Chu Kong Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ECKIRB1051203
Record Dates: First submitted 2018-05-08; First posted 2018-05-22 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Overactive Bladder Syndrome

STUDY DESIGN:
Intervention Model Description: overactive bladder patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- herbal patch group (Experimental): using herbal patch as an intervention
  Interventions: Drug: herbal patch
- placebo patch group (Placebo Comparator): using placebo patch as an intervention
  Interventions: Drug: placebo patch

INTERVENTIONS:
Drug: herbal patch — One patch with medicine should be applied to the skin every other day within two weeks
  Other Names: OAB patch
  Arms: herbal patch group
Drug: placebo patch — One patch without medicine should be applied to the skin every other day within two weeks
  Other Names: control patch
  Arms: placebo patch group

SUMMARY:
Overactive bladder is a clinical syndrome characterized by frequency, with or without urge incontinence, urgency, and nocturia, which affect patients' sleeping quality and rehabilitation program progressing. Current treatments include behavioral therapy (eg, life style adjustment, bladder training, pelvic floor muscle therapy) and medication. Antimuscarinic agents is the most common medications prescribed for OAB, but patients often have side effects like dry mouth and constipation. And there were plenty of herbal medicine which are beneficial to urine frequency and voiding dysfunction in ancient Chinese medicine books and records. In human trial, 62 Subjects diagnosed as overactive bladder will be enrolled and treated with Cinnamon patch. After treatment we will estimate the efficacy and record adverse events to conduct statistically analysis.

DETAILED DESCRIPTION:
Overactive bladder is a clinical syndrome characterized by frequency, with or without urge incontinence, urgency, and nocturia, which affect patients' sleeping quality and rehabilitation program progressing. Current treatments include behavioral therapy (eg, life style adjustment, bladder training, pelvic floor muscle therapy) and medication. Antimuscarinic agents is the most common medications prescribed for OAB, but patients often have side effects like dry mouth and constipation. And there were plenty of herbal medicine which are beneficial to urine frequency and voiding dysfunction in ancient Chinese medicine books and records. In human trial, 62 Subjects diagnosed as overactive bladder will be enrolled and treated with Cinnamon patch. After treatment we will estimate the efficacy and record adverse events to conduct statistically analysis.

The 1st year project: (1) Expect to enroll 62 clinical subjects of OAB. (2) Evaluate subjects 'symptom and proceed patch treatment. (3) Record treatment responses including adverse effect. (4) Conduct statistically analysis.

The 2nd year project: (1) Completing enrollment of 62 clinical subjects of OAB. (2) Finish evaluation and treatment of all subjects. (3) Statistically analysis all collecting data (4) Discuss and analyze the outcome.

ELIGIBILITY:
Inclusion Criteria:

* urgency score of OABSS ≥ 2 or total score of OABSS ≥ 3

Exclusion Criteria:

* suffering from acute urinary tract infection
* recurrent urinary tract infection ≥ 5 times in the last year
* Hematuria or bladder stone disease
* using foley catheter
* Pregnant or breastfeeding women
* Spinal cord injury patients
* Mental illness or substance abuse
* taking medicine for the treatment of overactive bladder within one month

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
OABSS | Change from Baseline OABSS at 2weeks
  Overactive bladder symptom score, questionnaire

SECONDARY OUTCOMES:
PPBC | Change from Baseline PPBC at 2weeks
  Patient perception of bladder condition, questionnaire
USS | Change from Baseline USS at 2weeks
  Urgency Severity Scale, questionnaire
TCMBCQ | Change from Baseline TCMBCQ at 2weeks
  Traditional Chinese Medicine Body Constitution Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: LIH-LIAN CHEN, MD, Principal Investigator — attending physician of department of Traditional Chinese medicine
Locations (1):
- EnChuKong hospital, New Taipei City, Sanxia Dist, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
primary and secondary outcome of this study
Supporting Information: ICF, CSR
Time Frame: information sharing after paper published
Access Criteria: all in public, without any kind of review